CLINICAL TRIAL: NCT02537197
Title: The Effect of Regular Naltrexone Dosing on Disordered Gamblers: An Examination of Neural Activation, Gambling Urges, and Gambling Behaviour
Brief Title: The Effect of Regular Naltrexone Dosing on Disordered Gamblers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Darren Robert Christensen, Principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB15-2025
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Gambling
MeSH Terms: conditions — Gambling | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Pre-post design, single treatment group
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Group (Experimental): Regular Naltrexone dosing (approximately 12 weeks): Initially, participants will be given seven 25mg oral naltrexone (ReVia, Generic Health, or similar) half tablets at intake (days 1-7). The Full dosing regimen will begin if no toxicity issues are present and consists of fourteen 50mg tablets (two per day; 100mg). If required, dosages can be stepped up or down. If adverse symptoms persist (or if gambling symptoms escalates), the participant will be removed from the study and given alternative treatments. Participants will receive the following week's medication at each Calgary Opioid Dependence Program visit. Pill counts will be made at each visit. Physicians will monitor the progress of participants from intake and adjust dosages up or down to control gambling behaviour.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Regular opioid antagonist dosing of disordered gamblers
  Other Names: Revia

SUMMARY:
This study examines the effect of regular naltrexone dosing on disordered gamblers. Gamblers will also be scanned pre- and post-treatment where we will investigate the functional changes to tasks designed to engage brain region associated with gambling and addiction. These changes will be correlated with treatment outcomes and urge scores.

DETAILED DESCRIPTION:
This study will investigate the effects of regular dosing of naltrexone for the treatment of disordered gambling. It will also examine the changes of neurological functioning to tasks associated with addiction. Converging evidence suggests that disordered gambling shares similarities with substance dependence and disordered alcohol use. Naltrexone is a medication that is used to reduce the cravings and euphoria from opioids and alcohol use and some studies have shown that it also has efficacy as a treatment for problematic gambling. Pilot data suggest the prefrontal cortex is activated for a healthy subject during a delay-discounting task, possibly indicating some consideration of the delayed value of a hypothetical money amount. If discounting rates can be correlated with treatment outcomes and neurological activation, these tasks may provide a new predictive tool for treatment outcome. However, no previous study has examined the neurological changes from pharmacological treatments of gambling. This study will provide data on the differences between pre- and post-treatment of regular naltrexone dosing for disordered gamblers

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age.
* Provide written consent.
* Evidence of Disordered Gambling (DSM-V; American Psychiatric Association, 2013)
* Seeking treatment for disordered gambling, referrals, or responding to information about the study presented in the media.
* Primarily Video Lottery Terminal gamblers (to standardize gamblers and as we are using stimuli in the gambling stimuli task that is similar to video lottery terminals displays so gamblers will be familiar with these images).
* Attendance at Alberta Health Service Evening Gambling Intensive Program (EGRIP) or similar
* English speaking

Exclusion Criteria:

* Evidence of a current significant medical illness, or unmanaged psychiatric or neurological disorder.
* Positive urine specimen to drugs of abuse.
* History of a traumatic brain injury or loss of consciousness (10 minutes or more).
* History of evidence of claustrophobia
* Left handed.
* Any condition or circumstance that prohibit imaging sessions such as metal implants.
* Contraindications to clinical doses of naltrexone.
* History or evidence of allergic reactions to naltrexone administration (i.e., rash, itching/swelling, severe dizziness, or trouble breathing).
* Concurrent use of additional alcohol dependence medication e.g. disulfiram.
* Evidence of current illicit opioid use
* Use of medications containing opioids/opiates
* Uncorrected visual impairment
* Evidence of brain abnormalities from structural scans
* Evidence of heart, liver or kidney failure.
* Failure to attend weekly EGRIP counselling sessions or similar
* Pregnant

Other Requirements:

* If sexually active must use contraception
* Cannot make ovum or sperm donation during study and six-months thereafter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04; Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Abstinence | 10-14 weeks
  No self reports of gambling

CONTACTS AND LOCATIONS:
Overall Officials: Darren R Christensen, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- Opioid Dependency Program, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No